CLINICAL TRIAL: NCT03181828
Title: Manipulating the Gut Microbiome Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The incidence of AEs was higher than the IB reported.
Sponsor: Nicholas Ah Mew (Other)
Responsible Party: Sponsor-Investigator, Nicholas Ah Mew, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: #7230; NCT02670889 (obsolete NCT alias)
Record Dates: First submitted 2017-06-01; First posted 2017-06-09 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Urea Cycle Disorder
Keywords: CPSI deficiency; OTC Deficiency; AS Deficiency; AL Deficiency
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Ornithine Carbamoyltransferase Deficiency Disease | interventions — acetohydroxamic acid

STUDY DESIGN:
Intervention Model Description: This pilot randomized crossover study will first evaluate the impact of AHA versus non-AHA primarily on intestinal flora cleavage of an infused bolus of 13C-Urea and secondarily on other biomarkers in healthy adults before applying the same crossover design to UCD subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acetohydroxamic Acid Oral Tablet then No Intervention (Experimental): Participants receive a single oral dose of 60 mg/kg acetohydroxamic acid (rounded to the nearest 250 mg) in the fasted state on the morning of the study. After completion of the 4-h study, participants then enter a wash-out period of 3 days. Participants then completed an identical 4-h study in the fasted state without acetohydroxamic acid.
  Interventions: Drug: Acetohydroxamic Acid Oral Tablet; Other: No treatment
- No Intervention then Acetohydroxamic Acid Oral Tablet (Experimental): Participants completed a 4-h study in the fasted state without acetohydroxamic acid. 3 days later, participants then completed an identical 4-h study in the fasted state, after having received a single oral dose of 60 mg/kg acetohydroxamic acid (rounded to the nearest 250 mg).
  Interventions: Drug: Acetohydroxamic Acid Oral Tablet; Other: No treatment

INTERVENTIONS:
Drug: Acetohydroxamic Acid Oral Tablet — A single oral dose of 60 mg/kg acetohydroxamic acid rounded to the nearest 250 mg tablet.
  Other Names: Lithostat
Other: No treatment — No treatment

SUMMARY:
The objective is to determine if acetohydroxamic acid (AHA) can prevent hydrolysis of urea by inhibiting the bacterial urease of gut flora of both healthy control adults as well as adults with urea cycle disorders

DETAILED DESCRIPTION:
This project will study the efficacy and safety of the pharmacologic blockade of urease in the nitrogen salvage pathway of intestinal microbes in subjects with partial urea cycle disorders. Additional trapping of ammonia as excretable urea may result in improved nitrogen excretion and reduced ammonia levels.

Urea cycle disorders (UCDs) are a group of disorders resulting from a complete or partial deficiency of one of the 6 enzymes or 2 transporters that comprise the urea cycle, the essential biochemical pathway which converts toxic ammonia into urea. These disorders have as a common feature, a reduced or complete inability to convert ammonia into urea, thereby resulting in high ammonia levels, or hyperammonemia. If untreated, hyperammonemia may result acutely in lethargy and coma, and chronically in intellectual disability. Current treatment for hyperammonemia is suboptimal, thus the search for new treatments is critical.

The urease inhibitor, acetohydroxamic acid (AHA, Lithostat®, Mission Pharmacal), is an FDA-approved product for another indication- the treatment of struvite nephrolithiasis in chronic urinary tract infections in both adults and children.

It is known that many urea-splitting bacteria also exist in the gut, and that in healthy individuals, approximately 15-30% of blood urea is degraded via gut bacteria into ammonia3, which returns to the liver via the portal vein, only to be recycled into urea. This percentage of degraded urea may even be greater in patients with urea cycle disorders, who are on a low protein-diet4 and whose gastrointestinal contents thus likely have lower nitrogen content, promoting bacterial recycling of nitrogen from available urea. Additionally, urea hydrolysis has been shown to be greatest in infants5, precisely the age at which hyperammonemic episodes are the most frequent in UCD patients.

We intend to study if AHA can inhibit gut bacteria degradation of urea, thereby reducing the quantity of ammonia returning to the liver. We intend to investigate this by studying subjects on two occasions at least 3 days apart:

On the first occasion, subjects will receive an intravenous dose of 13C-urea. Following the intravenous bolus of 13C-urea, over the subsequent 4 hours, we will collect several sequential measurements of blood and urine biomarkers from an IV catheter placed in the other arm. The intent is to obtain baseline 13CO2 kinetics in the subject.

On the second occasion, subjects will first receive an oral dose of AHA approximately 1 hour prior to the intravenous 13C-urea dose. Similar sequential measurements of blood and urine biomarkers will be performed. The intent is to observe a reduction in 13CO2 when AHA is administered.

We intend to initially study a cohort of unaffected adult subjects. If successful, we will study adults with partial urea cycle disorders.

This study will be conducted in the Clinical Research Center (CRC) of the Clinical and Translational Research Institute (CTSI) of Children's National Medical Center (CNMC).

ELIGIBILITY:
Inclusion Criteria:

* For Group 1 (healthy adults):
* Ages 18-60 years
* Compliant with receiving medications orally and intravenously
* Compliant with providing blood and urine samples

For Group 2 (adult UCD patients):

* Ages 18-60 years
* Compliant with receiving medications orally and intravenously
* Compliant with providing blood and urine samples
* Established diagnosis of CPSD, OTCD, ASSD or ASLD as follows:

  * Diagnosis of CPS I deficiency, defined as decreased (less than 20 % of control) CPS I enzyme activity in liver or an identified pathogenic mutation
  * Diagnosis of OTC deficiency, defined as the identification of a pathogenic mutation, linkage analysis in an affected family, less than 20% of control of OTC activity in the liver, or elevated urinary orotate (greater than 20 uM/mM) in a random sample or following allopurinol loading with absence of argininosuccinic acid
  * Diagnosis of AS deficiency (Citrullinemia), defined as a greater than or equal to 10-fold elevation of citrulline in plasma, decreased AS enzyme activity in cultured skin fibroblasts or other appropriate tissue, or identification of a pathogenic mutation in the AS gene
  * Diagnosis of AL deficiency (Argininosuccinic Aciduria, ASA), defined as the presence of argininosuccinic acid in the blood or urine, decreased AL enzyme activity in cultured skin fibroblasts or other appropriate tissue, or identification of a pathogenic mutation in the AL gene

Exclusion Criteria:

* For both Group 1 and Group 2:
* Current or prior Helicobacter pylori infection
* Chronic gastrointestinal illness (e.g., inflammatory bowel disease)
* Chronic renal failure
* Taking probiotic medications within a week of study start date
* Currently pregnant or lactating. Documentation of a negative pregnancy test within a week prior to testing is required, unless pre-menarchal or menopausal, experiencing menses that week, or other circumstances which preclude pregnancy (e.g. hysterectomy).
* Presence of acute infection at the time of inclusion
* Participation in any other clinical interventional trial or received experimental medication within the last 30 days
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at an additional risk by participating in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ah Mew, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- No Intervention, Then Acetohydroxamic Acid Oral Tablet [Lithostat]: Cross over from No Intervention- Non AHA; Period 1. Subjects (healthy adults and UCD patients) will receive a single oral dose of 60 mg/kg acetohydroxamic acid during one of the treatment periods, based on the randomization assignment determining whether treatment occurs in the first or the second treatment cycle; doses will be rounded to the nearest 250 mg to coincide with the available dosage form since the tablets cannot be scored.
- Acetohydroxamic Acid Oral Tablet [Lithostat], Then No Intervention: All subjects (healthy adults and UCD patients) will receive a single oral dose of 60 mg/kg acetohydroxamic acid during one of the treatment periods, based on the randomization assignment determining whether treatment occurs in the first or the second treatment cycle; doses will be rounded to the nearest 250 mg to coincide with the available dosage form since the tablets cannot be scored. Patients will be instructed to fast for 4 hours prior to the study; subsequently, the 13C-Urea tracer will be administered 60 minutes after the ingestion of the acetohydroxamic acid dose.
  Acetohydroxamic Acid Oral Tablet [Lithostat]: AHA:
  Acetohydroxamic acid has been an FDA approved medication for the treatment of struvite nephrolithiasis for over 25 years. According to the prescribing information, about 150 patients, including children, have been treated, most for periods of more than 1 year.
Period: Overall Study
Arm/Group | No Intervention, Then Acetohydroxamic Acid Oral Tablet [Lithostat] | Acetohydroxamic Acid Oral Tablet [Lithostat], Then No Intervention
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All the enrolled participants have been healthy adults.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention Then Acetohydroxamic Acid Oral Tablet | Acetohydroxamic Acid Oral Tablet Then No Intervention | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 47 [36 to 58] | 40 [38 to 42] | 43.5 [36 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Atom Percent Excess of 13CO2
Description: Difference in the % enrichment of Carbon-13 in blood CO2 as compared to baseline measurement, at sequential time points, after a single bolus of intravenous [13C]-Urea,
Time Frame: Time +0 minutes, +30 minutes, +60 minutes, +90 minutes, +120 minutes, +180 minutes, and +240 minutes from time of infused [13C] Urea IV
Measure: Mean (Standard Deviation); unit: Atom % Excess
Groups:
- Acetohydroxamic Acid Oral Tablet: Participants receive a single oral dose of 60 mg/kg acetohydroxamic acid (rounded to the nearest 250 mg) in the fasted state on the morning of the study.
- No Intervention: Participants completed a 4-h study in the fasted state without acetohydroxamic acid.
Arm/Group | Acetohydroxamic Acid Oral Tablet | No Intervention
Number analyzed (Participants) | 4 | 4
Atom % Excess
  0 min | 0 (0) | 0 (0)
  30 min | -0.00216 (0.00376) | 0.00268 (0.00531)
  60 min | 0.000959 (0.00130) | 0.000318 (0.0105)
  90 min | 0.00129 (0.00101) | 0.00336 (0.00583)
  120 min | 0.00152 (0.00117) | 0.00277 (0.00528)
  180 | -0.00392 (0.00561) | -0.000982 (0.00122)
  240 | -0.000537 (0.00386) | 0.00203 (0.00617)

2. Secondary Outcome: Blood [13C]-Urea
Description: Concentration of urea labeled with Carbon-13
Time Frame: Time +O minutes, +30 minutes, +60 minutes, +90 minutes, +120 minutes, +180 minutes, and +240 minutes from time of [13C] Urea IV
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Acetohydroxamic Acid Oral Tablet | No Intervention
Number analyzed (Participants) | 4 | 4
micromol/L
  0 Min | 0 (0) | 0 (0)
  30 Min | 174.9 (43.57) | 199.5 (9.12)
  60 Min | 151.9 (30.05) | 165.2 (6.07)
  90 Min | 140.9 (12.48) | 152.4 (6.14)
  120 Min | 137.3 (9.58) | 136.8 (6.65)
  180 Min | 127.8 (9.87) | 126.5 (7.78)
  240 | 119.9 (11.93) | 117.2 (9.95)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Acetohydroxamic Acid Oral Tablet | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetohydroxamic Acid Oral Tablet (N=4) | No Intervention (N=4)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Nausea (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03181828/Prot_SAP_ICF_001.pdf